CLINICAL TRIAL: NCT03868436
Title: A Phase IV Real World Study on the Use of Low Dose Methoxyflurane (PENTHROX™) for the Treatment of Moderate to Severe Trauma Pain in the Canadian Emergency Department
Brief Title: PENTHROX™ in the Canadian Emergency Department (ED)
Acronym: ADVANCE-ED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Purdue Pharma, Canada (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN-MEOF-MA-OO1
Record Dates: First submitted 2019-02-21; First posted 2019-03-11 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Methoxyflurane

STUDY DESIGN:
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methoxyflurane (MEOF)-active treatment (Other): single arm study all subjects will be treated with Methoxyflurane 3 mL
  Interventions: Drug: Methoxyflurane 3mL

INTERVENTIONS:
Drug: Methoxyflurane 3mL — As soon as possible following enrollment and initial procedures, the patient will be supplied with a PENTHROX™ kit which includes one inhaler containing 3 mL of MEOF for pain management. A member of the research team will train the patient to self-administer MEOF. PENTHROX™ is an approved (trademarked) product in Canada and is commercially available in a combination blister pack with one 3 mL sealed bottle and one PENTHROX™ inhaler with the Activated Carbon (AC) chamber.
  Other Names: PENTHROX™

SUMMARY:
This Canadian, multi-centre, prospective, real world study is designed to evaluate the effectiveness of low dose methoxyflurane (MEOF) (PENTHROX™) for the treatment of moderate to severe pain associated with trauma in the Canadian ED.

DETAILED DESCRIPTION:
The study will assess the change in pain intensity over 20 minutes from start of administration of PENTHROX™ and will generate Real World Evidence in support of existing clinical trial data including effectiveness, safety and additional parameters of low dose MEOF (PENTHROX™) in Canadian EDs.

ELIGIBILITY:
Inclusion Criteria:

1. Conscious adult patients: ≥ 18 years of age
2. Moderate to severe pain associated with trauma (NRS0-10 ≥ 4) which is unlikely to require surgery/hospitalization, such as

   * Musculoskeletal injuries and physical wounds
   * Fractures
   * Lacerations
   * Burns
   * Dislocations
   * Contusions
   * Injury due to foreign bodies
3. Patient (and/or patient's authorized legal representative) should understand the nature of the study and provide written informed consent
4. Patient is able to follow all study requirements and procedures and complete required questionnaires

Exclusion Criteria:

1. Multi-level trauma
2. Women of child bearing potential who are pregnant or peri partum, including labour
3. An altered level of consciousness, due to any cause, including head injury, drugs, or alcohol
4. Clinically significant renal impairment
5. A history of liver dysfunction after previous MEOF use or other halogenated anesthetics
6. Hypersensitivity to MEOF or other halogenated anesthetics, or to butylated hydroxytoluene
7. Known or genetically susceptible to malignant hyperthermia or a history of severe adverse reactions in either patient or relatives
8. Exacerbation of an underlying condition (i.e., chronic pain)
9. Clinically evident or potential hemodynamic instability as per the opinion of the investigator
10. Clinically evident respiratory impairment as per the opinion of the investigator
11. Prior treatment with PENTHROX within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Change in mean pain intensity: Numerical Rating Scale | 20 mins from start of administration (STA) of PENTHROX™
  The level of pain intensity will be collected by means of the Numerical Rating Scale (NRS). The NRS is considered a reliable and valid scale for assessing pain intensity and is preferred by patients for its simplicity. In this 11-point scale, the end points are the extremes of no pain and pain as bad as it could be, or worst pain (i.e. a score of 0 = no pain and a score of 10 = worst pain possible).
  Assessed by the patient 20 mins post PENTHROX™ inhalation

SECONDARY OUTCOMES:
Speed of action of analgesia | At any point from STA of PENTHROX™ to 20 mins post inhalation
  Speed of action of analgesia is defined as the time at which the patient experiences meaningful pain relief following inhalation of PENTHROX™.
  The healthcare professional will instruct the patient to note the time at which they experience meaningful pain relief. The time point will be recorded in the case report form.
Proportion of treatment-emergent adverse events (TEAEs) | At any point From STA of PENTHROX™ until the end of the observation period (24 hours)
  Assessment of patient reported adverse events throughout the observation period.
Global Medication Performance (GMP) before discharge from ED (Patient & Health Care Professional) | at 20 minutes From STA of PENTHROX™ and at the end of the observation period (up to 24hours)
  Global medication performance (GMP) is an assessment of the health care professional's and patient's impression of how well a medication works.
  Global Medication Performance (GMP)-is a patient and health care provider reported outcome with the objective of assessing the health care professional's and patient's impression of how well a medication works.
  GMP is measured by asking the patient and health care professional a single question: "rate the pain relief provided by PENTHROX™" utilizing a 5-point Likert scale where 1=Poor- 5=Excellent
Fulfillment of pain relief expectations (Patient & Healthcare professional) | At the end of the observation period (up to 24hours)
  Fulfillment of pain relief expectations- is a patient and health care professional reported outcome with the objective of assessing the health care professional's and patient's impression of how well a medication fulfilled their expectations.
  Fulfillment of pain relief expectations is measured by asking the patient and health care professional a single question: "To what extent has your expectations regarding pain control been met" and utilizing a 5-point Likert scale where 1=Poor- 5=Excellent.
Use of rescue medication | From STA of PENTHROX™ to the end of the observation period (up to 24hours)
  The time of first use of rescue medication after STA of PENTHROX™ up to and including 60 minutes will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Dhani, PhD, Study Director — Purdue Pharma, Canada
Locations (6):
- Canada (6):
  - Charles V Keating Emergency and Trauma Centre, QEII, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Markham Stouffville, Markham, Ontario
  - St. Joseph's Healthcare, Welland, Ontario
  - Centre Integre Universitaire De Sante Et De Service Sociaux (CIUSSS) Saguenay-Lac-Saint Jean, Chicoutimi, Quebec
  - Centre Intégré de Santé et de Services Sociaux de la Montérégie-Centre, Greenfield Park, Quebec

IPD SHARING:
Plan to Share IPD: No